CLINICAL TRIAL: NCT06628648
Title: Hypertension as a Reason for Concellation of Elective Minor Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: University Tunis El Manar (Other)
Responsible Party: Principal Investigator, HibetAllah Ktata, associate Professor, University Tunis El Manar
Other Study IDs: UTEM HCS
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Hypertension Secondary; Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- canceled: Hypertensive patients proposed for minor abdominal surgery and canceled for high blood pressure numbers.
- not canceled: Hypertensive patients proposed for minor abdominal surgery not canceled: whose blood pressure figures are correct.

SUMMARY:
During the anesthesia outpatient consultation, patients proposed for minor abdominal surgery, known hypertensive patients are selected.

On the day of the procedure, we check the blood pressure figures. If the numbers are high: SBP ≥ 180 and/or PAD≥110: we start by a filling as well as a dose of 1 mg Midazolam IV and the blood pressure figures are re-evaluated. If 3 measurements blood pressure figures remain above the threshold values: Surgery is postponed and the patient will be included to group (A) for canceled. If the blood pressure figures are correct, the surgery is accepted and the patient will be included in the group (NA) for not canceled.

DETAILED DESCRIPTION:
During the anesthesia outpatient consultation, patients proposed for minor abdominal surgery, known hypertensive patients are selected. If the blood pressure figures are balanced in the previous 12 months, they are included in the study and the anesthesiologist informs them of the study protocol and obtains their consent.

On the day of the procedure, the patient is admitted to the operating room. We begin warming the patient and carry out standard monitoring, then, we check the blood pressure figures. If the numbers are high: SBP ≥ 180 and/or PAD≥110: we start by a filling as well as a dose of 1 mg Midazolam IV and the blood pressure figures are re-evaluated. If 3 measurements blood pressure figures remain above the threshold values: Surgery is postponed and the patient will be included to group (A) for canceled. If the blood pressure figures are correct, the surgery is accepted and the patient will be included in the group (NA) for not canceled.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or over, consenting
* known hypertensive patients.
* Patients proposed for planned minor abdominal surgery (≤ 2 hours).

Exclusion Criteria:

* patients not premedicated (antihypertensive treatment)

Non-inclusion criteria:

* patient refusal .history of hypertensive emergency within 06 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included for this study: proposed for minor abdominal surgery, known hypertensive, prepared for the surgical procedure. Patient recruitment will be carried out over a period of 7 months by the anesthesia team with cooperation from the general surgery team.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-15 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
Incidence of surgery canceled due to high blood pressure figures in the operating room. | In the operating room
  In the operating room, if the blood pressure figures are high(according to BHS recommendations from 2016) the surgery is canceled

SECONDARY OUTCOMES:
Score d'anxiété: Amsterdam Preoperative Anxiety and Information Scale (APAIS) | before entering the operating room
  The APAIS scale is presented in the form of a questionnaire composed of six questions, the first three of which assess the patient's anxiety relating to anesthesia, the following two assess the patient's anxiety relating to surgery, and finally a last question assesses the patient's desire for information.
  The minimum score is 6 and the maximum is 20. If the score is greater than 11, this means that the patient's level of anxiety is high
The quality of reception in the operating room | before entering the operating room
  Patient satisfaction: Bad/average/good
History of cancellation for hypertension in the operating room | Pre-operative, at the anesthesia consultation
  presence or absence of a history of cancellation for high blood pressure figures
specify the anti-hypertension molecule | Pre-operative, at the anesthesia consultation
  the antihypertensive molecule taken by the patient as background treatment
Control and monitoring of hypertension Control and monitoring of hypertension Control and monitoring of hypertension | During the pre-anesthesia consultation
  The patient is followed-up in town: by a general practitioner or a cardiologist
Entrance to the operating room: on foot, chair or trolley | before entering the operating room
  Arrival at the operating room: on foot, chair or trolley
Day of the week | before entering the operating room
  Day of the week: from Monday to Saturday
Waiting time before entering the operating room (in minutes) | before entering the operating room
  waiting time before entering the operating room: in minutes

CONTACTS AND LOCATIONS:
Overall Officials: BENALI MECHAAL, Professor, Principal Investigator — maamouri nabeul
Locations (1):
- HIBET ALLAH ktata, Nabeul, Tunisia